CLINICAL TRIAL: NCT05941013
Title: Ultrasound-detectable Endotracheal Tube: a Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: John R. Charpie (Other)
Responsible Party: Sponsor-Investigator, John R. Charpie, Professor of Pediatric Cardiology, Professor of Pediatrics, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HUM00234901
Record Dates: First submitted 2023-05-31; First posted 2023-07-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cardiac Catheterization; Endotracheal Tube
Keywords: Ultrasound; Intubation

STUDY DESIGN:
Masking Description: The outcomes assessor is "blinded" for outcome measure 4. Specifically the protocol says, "After each case is completed, the fluoroscopic images and ultrasound images will be interpreted by independent study team members who are blinded to the results of the other test."
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Ultrasound detectable cuffed endotracheal tube (USD-ETT) (Experimental): Intubation with a novel ultrasound-detectable endotracheal tube
  Interventions: Device: Ultrasound detectable cuffed endotracheal tube (USD-ETT)

INTERVENTIONS:
Device: Ultrasound detectable cuffed endotracheal tube (USD-ETT) — Intubation with a novel ultrasound-detectable endotracheal tube

SUMMARY:
The researchers are studying whether special features make it easier to see if the breathing tube is in the correct place. It is hoped that the investigational device will enable more accurate placement (depth and trachea vs. esophagus).

DETAILED DESCRIPTION:
The participant will have a breathing tube where the balloon (cuff) at the end of the tube has two special features: 1) The balloon will have a divot in it, rather than be round in shape, and 2) The balloon will be filled with saline (salt water), rather than air. The breathing tube is called an ultrasound detectable cuffed endotracheal tube (USD-ETT).

The USD-ETT has not been tested or used in humans previously.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing scheduled or planned diagnostic or interventional cardiac catheterization with planned general anesthesia requiring endotracheal intubation.

Exclusion Criteria:

* Patient has a known airway abnormality, including tracheal stenosis, previous tracheal stenosis, or tracheobronchomalacia.
* Patient has a tracheostomy.
* Patient is ventilator-dependent.
* Patient has an anticipated difficult intubation based upon airway exam and/or history of difficult intubation.
* Patient is unlikely (in opinion of anesthesia team) or is unable to be intubated with 3.5 mm, 4.0 mm, or 4.5 mm Inner Diameter USD-ETT due to the size of the patient or their airway.
* Patient is already intubated prior to the scheduled procedure.
* It is anticipated that the patient will not be extubated after the catheterization procedure.
* Concurrent enrollment in another clinical trial with an intervention during the cardiac catheterization procedure or 30 days afterwards.
* Allergy to plastic/materials in USD-ETT

Ages: 6 Months to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of the USD-ETTs visualized by ultrasound | Within 5 minutes of placing the ultrasound probe at the suprasternal notch after intubation
  Reported as a 'yes' or 'no' - this outcome simply seeks to verify if the ultrasound can detect the ultrasound detectable cuffed endotracheal tube. The outcome measure assesses if the device is detectable as designed. It does not assess health related information.

SECONDARY OUTCOMES:
Adverse events that could be related to the USD-ETT device | Up to 30 days post intubation
Safely support ventilation and oxygenation of the patient during the procedure | Immediately following extubation
  Assessed by the question: "Were there any desaturation events, inability to property ventilate the patient or, blood gas abnormalities, that could be attributable to the ETT?" will be described
Kappa agreement between placement location of USD-ETT as assessed by ultrasound and fluoroscopy | Approximately 5 minutes after of placing the ultrasound probe at the suprasternal notch after intubation
  Ultrasound location data compared to fluoroscopy location data using a weighted Kappa statistic

CONTACTS AND LOCATIONS:
Overall Officials: John Charpie, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No